CLINICAL TRIAL: NCT00006443
Title: Evaluating Responses to Antiretroviral Drugs in Cells and Tissues (The ERADICATE Study): Comprehensive Comparisons of Viral and Cellular Dynamics Among Previously-Untreated Subjects With Acute HIV Infection (Seroconversion Syndrome) or Recently Acquired HIV Infection Versus the Early, Middle, and Advanced Stages of Seropositive HIV Infection
Brief Title: Effectiveness of Anti-HIV Drugs in Patients Who Have Not Received Previous Anti-HIV Drugs During Different Stages of HIV Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Purpose: Treatment
Other Study IDs: AIEDRP AI-08-002; PHA 082
Record Dates: First submitted 2000-11-03; First posted 2001-08-31 (Estimated); Last update posted 2011-03-02 (Estimated); Status verified 2005-01

CONDITIONS: HIV Infections
Keywords: T-Lymphocytes; HIV-1; Lymphoid Tissue; Stavudine; HIV Protease Inhibitors; Polymerase Chain Reaction; Biological Markers; Lamivudine; Indinavir; RNA, Viral; Genotype; Phenotype; Cytokines; Nelfinavir; Macrophages; Reverse Transcriptase Inhibitors; In Situ Hybridization; Anti-HIV Agents; Viral Load; Cell Membrane; Acute Infection; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; Nelfinavir; Lamivudine; Stavudine

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Nelfinavir mesylate
Drug: Lamivudine
Drug: Stavudine

SUMMARY:
The purpose of this study is to compare changes in HIV levels and certain immune cells among patients at different stages of HIV infection. This study will also see how a combination of stavudine (d4T), lamivudine (3TC), indinavir (IDV), and nelfinavir (NFV) affects these levels.

Current findings in anti-HIV drug treatment have led to a greater understanding of the background of HIV. To find the best anti-HIV treatment to eliminate all HIV viruses, cells and tissues infected with the HIV virus are examined after combination anti-HIV treatment, when the level of HIV infection is low. The ERADICATE study will examine the idea that HIV viruses can be eliminated at any stage of infection over time.

DETAILED DESCRIPTION:
Recent advancements in antiretroviral therapy have led to a better understanding of the natural history and immunopathogenesis of HIV-1 infection. To calculate the degree and duration of antiretroviral effect necessary to eliminate infection, characterization of residual cellular and tissue HIV reservoirs following high-level viral suppression is necessary. The ERADICATE study will evaluate the hypothesis that complete viral inhibition is possible, regardless of HIV disease stage, and leads to HIV eradication from tissues over time.

Patients are divided into 1 of 5 groups based on the stage of HIV infection. Patients receive oral stavudine (d4T), lamivudine (3TC), indinavir (IDV), and nelfinavir (NFV) twice daily for 24 weeks. All patients undergo basic blood sampling to follow HIV-1 RNA levels and absolute T cell subset numbers daily for 5 days; then 3 times a week for 3 weeks; 2 times a week for 4 weeks; every 2 weeks for 12 weeks; and monthly thereafter for a total of 3 years. In addition, the following tissues are sampled at baseline and after 2 weeks and 6 months on therapy: 1) lymph node; 2) tonsillar; 3) perirectal lymphoid; 4) cerebrospinal fluid; 5) and semen.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are infected with HIV and have had certain tests to indicate the stage of their disease.
* Are at least 18 years old.
* Practice birth control during the study.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have received anti-HIV medication for more than 1 week.
* Have a serious AIDS-related infection or other illness.
* Require medication that interferes with the study drugs.
* Have had a peripheral neuropathy, a painful condition affecting the nervous system.
* Have been given drugs that affect the immune system within 2 weeks before study entry.
* Have a bleeding disorder including hemophilia.
* Abuse alcohol or substances.
* Are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Primary Completion 2003-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Michael S. Saag, Birmingham, Alabama, United States